CLINICAL TRIAL: NCT00353236
Title: The Contribution of Internal Maternal Resources to Creation of Motherhood. Comparison Among Mothers to Twins and Singleton
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Other Study IDs: SHEBA-06-4170-JK-CTIL
Record Dates: First submitted 2006-07-17; First posted 2006-07-18 (Estimated); Last update posted 2006-07-18 (Estimated); Status verified 2006-07

CONDITIONS: Preterm Birth
Keywords: delivery of preterm infant and/or twins
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

SUMMARY:
Delivery of twins or preterm infant is a very stressful episode to mothers. The purpose of this study is to characterize maternal psychological resources in dealing with this situation and compare it to mothers giving birth to singleton at term

ELIGIBILITY:
Inclusion Criteria:

* Study group: Mothers who give birth to twins or preterm infants
* Control: Mothers who give birth to singleton, full term infants

Exclusion Criteria:

* None

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Kuint, MD, Study Director — Sheba Medical Center
Locations (1):
- Sheba Medical Center - Neonatal Department, Ramat Gan, Israel